CLINICAL TRIAL: NCT02437552
Title: Cycle Ergometer Exercise in Phase I of Cardiac Rehabilitation After Cardiac Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study would be conducted by a master course student, nevertheless, she was unable to go forward with it.
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ada Clarice Gastaldi, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USP 2015-1
Record Dates: First submitted 2015-04-29; First posted 2015-05-07 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Exercise Movement Techniques; Cardiac Surgery
Keywords: Cardiac Surgery, Coronary Artery Bypass, Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group: routine physiotherapy (Placebo Comparator): Are patients who carry out the routine already established the Unit, consisting of the first post surgery, the patient lying down doing the breathing exercises, active exercises ends and active-assisted upper (UL) and lower limbs (LL),
  Interventions: Other: routine physiotherapy
- Intervention group: ergometer cycle exercise (Active Comparator): Are the patients who will carry out the exercises routine over the cycle ergometer twice daily from 3 PO for 5 minutes with its progressiveness at discharge for ward for 10 minutes
  Interventions: Device: ergometer cycle exercise; Other: routine physiotherapy

INTERVENTIONS:
Device: ergometer cycle exercise
  Arms: Intervention group: ergometer cycle exercise
Other: routine physiotherapy — routine physiotherapy

SUMMARY:
The prevalence of heart diseases has increased significantly in recent years and it is a health public problem due to an increased risk of death by several reasons. A cardiac surgery is an alternative of treatment for critical injuries heart valves and coronaries arteries. Changes in respiratory system resulting from cardiac surgery are well established and include a reduced functional capacity due post-surgical pain, causing increased respiratory function and increased oxygen consumption . The exercises with the cycle ergometer in phase I of cardiac rehabilitation can improve peripheral muscle strength, functional capacity and perception of dyspnea when used postoperatively and there are speculations if an earlier carried out can contribute to a better postoperative evolution of patients, but these benefits in phase I of the Rehabilitation Cardiac are not well defined in the literature. Objective: To evaluate the exercises effects with ergometer cycle in the postoperative course of patients undergoing cardiac surgery. Method: Patients will be recruited the cardiac surgery service of Polyclinic Pato Branco in the city of Pato Branco in state of Paraná, of both sexes, appropriate for the inclusion criteria, which will be evaluated by pulmonary function tests (strength of respiratory muscles, submaximal exercise test, dyspnea scales, laboratories tests and radiological exam). All patients will be randomly assigned for one of two groups: the control group (Conventional treatment) and rehabilitation group (conventional treatment +cycle ergometer), for about 7 days at postoperative period. Patients will be reevaluated on the third postoperative day and at discharge. Clinical evolution data will be collected from the records and notes of the medical staff and monitoring physiotherapist.

DETAILED DESCRIPTION:
The research will be a randomized controlled clinical trial. The study will be conducted at the Polyclinic Pato Branco, in the city of Pato Branco Parana - Brazil and this study already approved by the Ethics Committee Clinical Hospital and Faculty of Medicine, University of São Paulo and all participants sign the consent form informed. For the implementation of research wil be recruited patients heart surgery who fit the inclusion criteria and do not show any characteristics of the exclusion criteria, which agree to participate and sign the consent form free and informed. The equipment and tests are already included in routine admissions of patients, approved by the hospital and the Brazilian Public Health System (SUS).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery type Myocardial Revascularization and Exchange Mitral Valve Aortic, both sexes and aged between 30-75 years.

Exclusion Criteria:

* Patients undergoing surgical correction of heart disease congenital, aortic aneurysm and dissection of aorta;

  * Present disabling disease to accomplish what is proposed in study as previous stroke, mental or motor deficit, hearing loss, amputation of the lower limbs (unilateral or bilateral);
  * Present psychomotor agitation of immediate postoperative and first postoperative and history weaning failure in the immediate;
  * Instability hemodynamics and vasoactive drugs;
  * Present what other type of peri and postoperative complications;
  * Re-operation within 24 hrs.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Change of six-minute walk test (6MMWT) distance | Before surgery ,third and seventh postoperative day
  The six-minute walk test will be conducted with monitoring blood pressure, HR, RR and SpO2 in a hall plan, with distances previously marked. The patient will be accompanied by the researcher and encouraged by constant verbal stimulation, walking as fast as possible, if the patient stop walking the timer will keep triggered. Will use the oximeter with the sensor on the third finger of the right hand, and a certain reading after the signal stabilization and at the same time we get the heart rate. Will be used to calculate the expected value, and reference to distance in the 6MWT, the equations proposed by Enright and Sherrill (1998) determining the percentage of predicted for each test performed by patient.

SECONDARY OUTCOMES:
Change of spirometric values | Before surgery ,third and seventh postoperative day
  Spirometry will be performed according to criteria of the American Thoracic Society and the Brazilian Consensus Spirometry. Values will be observed from CVF, VEF1 e PEF.

OTHER OUTCOMES:
Change of respiratory muscle strength - Mouth pressure measurements | Before surgery ,third and seventh postoperative day
  Manovacuometry will be performed with the patient seated with nasal clip, the display scale with intervals of 4 cmH2O and variation +/- 120 cmH2O. The highest value obtained during the two maneuvers will be compared to the table described by Neder et al (1999), which predicts expected values for the Brazilian population according to gender and age.
Change of perceived dyspnea | Before surgery ,third and seventh postoperative day
  The perceived effort is used the Borg Scale modified scored from 0 to 10. And dyspnea scale will be scored from 0 to 4 according to the intensity of dyspnea and is based on used the scale of the Medical Research Council (MRC).
Change of body mass index | Before surgery and postoperative seventh day
  The BMI will be calculated using the classical formula: BMI = current weight (kg) / A2 (m). The following lower limits of normal were considered: BMI <21 for age group 35-44 years; <22 for 45-54 years; <23 for 55 -64 years and <24 to 65 above years.
Change of cirtometry | Before surgery ,third and seventh posoperative day
  Cirtometry will be held in myocardial revascularization of patients who use the saphenous and waist hip will be performed in all patients. Will be used a tape measure.
Change of peripheral muscle strength | Before surgery ,third and seventh postoperative day
  The peripheral muscle strength assessment test will be the end of the test the foot, the patient will be instructed to stay barefoot with his right hand resting on the front wall and with a semi elbow flexion to aid maintenance balance. Prior to testing, the participant will be oriented make a plantar flexion to the point of support of the joints metatarsophalangeal and this time will be marked by the examiner through a mark on the wall and the patient will be informed that should reach the one marked point. The test itself consisted of time, in seconds, the time it takes to perform five push-ups as plantar soon as possible.
Change in cortisol levels | Before surgery ,third and seventh postoperative day
  Laboratory evaluation will be performed by laboratory staff of hospital with a blood sample from the patient, which will be assessed the cortisol levels .
change of radiological assessment | Before surgery ,third and seventh postoperative day
  Radiological assessment will be held the day before the surgery, the third post-operative and post-operative seventh, the clinic Radiology Southwest - Pato Branco - Paraná to assess complications lung from surgery.
Adherence evaluation | Third and seventh postoperative day
  The questionnaire will be administered at the end of the first contact of the patient the exercises with the cycle ergometer to assess adherence running a differential exercise during your surgical recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlínica Pato Branco, Pato Branco, Paraná, Brazil

REFERENCES:
- [Result] BAUMGARTEN, M.C.S. et al. Behavior of pain and pulmonary function in patients undergoing heart surgery via sternotomy. Rev Bras-surgical Cardiovasc.24 (4), 2009 BRUMMEL, N.S; GIRARD, T.D. Preventing delirium in the intensive care unit.Crit Care Clin. 29(1):51-65 , 2013. Guidelines on Cardiopulmonary and Metabolic Rehabilitation: Practical Aspects and Responsibilities. Arq Bras Cardiol of. V. 86, No. 1, January 2006. Available in http://publicacoes.cardiol.br/consenso/2006/8601012.pdf> access 10/14/14, 13h22min. ENRIGHT IP SHERRIL DI. Reference equations for the six minute walk in healthy adults. Am J Respir Crit Care Med. V.158, p.1384-1387,1998.